CLINICAL TRIAL: NCT02334410
Title: Early Intervention to Reduce Bone Loss After Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Strathclyde (Other)
Collaborators: Queen Elizabeth National Spinal Injuries Unit, Glasgow (Unknown)
Responsible Party: Principal Investigator, Sylvie Coupaud, Dr, University of Strathclyde
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UEC14/57
Record Dates: First submitted 2015-01-06; First posted 2015-01-08 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Spinal Cord Injury; Osteoporosis
Keywords: fractures; immobilisation; paraplegia; tetraplegia
MeSH Terms: conditions — Spinal Cord Injuries; Osteoporosis; Fractures, Bone; Paraplegia; Quadriplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reference (No Intervention)
- Whole body vibration (WBV) (Experimental): Vibration therapy
  Interventions: Device: Whole body vibration (WBV)

INTERVENTIONS:
Device: Whole body vibration (WBV) — Side-alternating WBV
  Other Names: Galileo (Novotec Medizintechnik)
  Arms: Whole body vibration (WBV)

SUMMARY:
After a complete spinal cord injury (SCI), the patient becomes wheelchair-dependent, and the associated lack of weight-bearing and inactivity of paralysed muscles can lead to extensive bone loss in the long bones of the legs. It has been documented that the most rapid phase of bone loss is during the first year, but bone loss can continue for a number of years post-injury, leading to an increased risk of fracture in chronic SCI. Through a previous longitudinal study, in which we described rates of bone loss in the first year of SCI using peripheral Quantitative Computed Tomography (pQCT), we showed that there is a subset of patients who suffer from extremely rapid bone loss, losing up to 50% of their bone mineral density (BMD) in the first 12 months post-SCI. As a result of this work, we now know that, by performing repeat bone scans within months of injury, we are able to detect and "red-flag" those patients at highest risk of rapidly weakening bones. We propose that, once these patients have been identified, there is an opportunity to intervene with bone-stimulating interventions within months of injury, before BMD reaches dangerously low values. In this new phase of the research, therefore, we are introducing an intervention phase to the longitudinal pQCT study. For this, we aim to trial a physical intervention, Whole Body Vibration (WBV), that could potentially reduce rates of further bone loss in fast bone losers. Vibration would achieve this by acting as a mechanical stimulus for bone cells, to encourage bone formation. If shown to be successful as an early bone-stimulating intervention, it may prove to be a tool for reducing future fracture risk in patients with SCI.

ELIGIBILITY:
Inclusion Criteria:

* Motor-complete spinal cord injury (SCI)
* SCI at neurological levels C4 and below
* Within six weeks of SCI

Exclusion Criteria:

* Recent bilateral fractures in tibia and/or femur
* Previously diagnosed osteoporosis
* Pregnancy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-02; Primary Completion 2018-01 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Rate of change of bone mineral density (BMD) based on peripheral Quantitative Computed Tomography (pQCT) bone scans | 12 months
  Can WBV intervention reduce the rate of bone loss in patients with early spinal cord injury?
Rate of change of calcium and bone profiles based on blood samples | 12 months
  Biochemical markers of bone formation, bone resorption, hormone and mineral levels.

SECONDARY OUTCOMES:
Correlation between imaging and biochemical markers of bone health | 12 months
  Imaging-derived data will be compared with analyses of blood samples as indicators of bone health

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Elizabeth National Spinal Injuries Unit, Glasgow, United Kingdom